CLINICAL TRIAL: NCT03709368
Title: Effect of Two add-on Software Interventions for Improving Hand Washing and Sanitation in Rural Tanzania: an Impact Evaluation
Brief Title: Software Interventions for Improving Hand Washing and Sanitation in Rural Tanzania: an Impact Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Evidence-Based Practice, Belgium (Other)
Collaborators: Tanzania Red Cross Society (Unknown); Muhimbili University of Health and Allied Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: TAN-001
Record Dates: First submitted 2018-10-02; First posted 2018-10-17 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Diarrhea
Keywords: Hand washing; WASH; RANAS; Behavior change
MeSH Terms: conditions — Diarrhea | interventions — Equipment and Supplies

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- RANAS (Experimental): Hardware CLTS+PHAST RANAS (contextualized)
  Interventions: Other: Hardware; Behavioral: CLTS; Behavioral: PHAST; Behavioral: RANAS
- Mini-RANAS (Experimental): Hardware CLTS+PHAST mini-RANAS (norms)
  Interventions: Other: Hardware; Behavioral: CLTS; Behavioral: PHAST; Behavioral: mini-RANAS
- Control (Active Comparator): Hardware CLTS+PHAST Placebo
  Interventions: Other: Hardware; Behavioral: CLTS; Behavioral: PHAST; Other: Placebo poster

INTERVENTIONS:
Other: Hardware — Community sessions will be provided to each of the sub-villages (n=27) teaching participants how to build a tippy tap, how to build an improved latrine, and how to make liquid soap. In addition, an existing water gravity flow scheme will be rehabilitated and extended, 350 tippy taps and 350 pans for pour flush latrines will be distributed, and sanitation blocks will be built in four schools. Within these schools, SWASH school hygiene clubs will be organized.
Behavioral: CLTS — CLTS sanitation and HW sessions will be given. A first session will focus on sanitation, covering 7 exercises: 1) sanitation or social map, 2) transect walk, 3) shit calculation, 4) medical expenses, 5) shit flow diagram, and 6) water/shit demo, 7) community declaration. A second session will focus on HW, involving 10 exercises: 1) anal cleansing materials, 2) shit and shake, 3) cassava/egg demonstration, 4) charcoal smearing, 5) smelly hands, 6) feces on baby nappies, 7) scratch & smell, 8) wall contamination, 9) food sharing, 10) dirt under fingernails. These sessions will take approximately 3-5 hours each. Follow-up community meetings and household visits will take place to monitor improvement.
Behavioral: PHAST — PHAST sessions are based on the 'PHAST step-by-step guide: A participatory approach for the control of diarrhoeal disease' of the World Health Organization. Considering the overlap with some CLTS activities, only a selection of the full guideline will be enrolled, namely: 1) Health problems in our community, 2) Good and bad hygiene behaviors, 3) Investigating community practices, 4) How diseases spread, 5) Blocking the spread of disease, 6) Selecting the barriers, 7) Choosing sanitation improvements, and 8) Choosing improved hygiene behaviors. These 8 activities will be enrolled in approximately 40 community groups. Each activity will take between 30 minutes - 2 hours to complete.
Behavioral: RANAS — Nine household visits of 20-40 min each will be offered at a frequency of one visit every two months. The content of these add-on visits is based on the RANAS manual: 'Systematic Behavior Change in Water, Sanitation and Hygiene - A practical guide to using the RANAS approach' (www.ranasmosler.com). First, baseline data is gathered through a questionnaire to better understand the context that is at play. Next, this data is analyzed in a do'er non-do'er analysis. Only those behavioral factors that are significantly different between do'ers and non-do'ers will be included in the intervention, as these are, at least theoretically, considered to be decisive for HW and latrine use behavior in the current setting.
  Arms: RANAS
Behavioral: mini-RANAS — Nine household visits of 20-40 min each will be offered at a frequency of one visit every two months. The content of the mini-RANAS add-on intervention is based on the 'Norm Behavior Change Techniques' from the RANAS manual 'Systematic Behavior Change in Water, Sanitation and Hygiene - A practical guide to using the RANAS approach' (www.ranasmosler.com). During the mini-RANAS household visits, emphasis will be put on norms and volunteers will encourage participants to become a role model by improving HW and sanitation infrastructure and behavior.
  Arms: Mini-RANAS
Other: Placebo poster — One household visit will be offered. During this visit, a placebo poster will be distributed focusing on first aid. The topics to be discussed are burns, cuts and grazes. The main goal of this household visit is to avoid jealousy among the control cohort.
  Arms: Control

SUMMARY:
BACKGROUND. Diarrhea is ubiquitous, particularly among people in low- and middle-income countries. Unsafe drinking water, poor sanitation, and insufficient hygiene are responsible for nearly 90% of diarrhea-related mortalities. Despite extensive knowledge that has been obtained in recent years, there is no consensus as to the most efficacious approach to improve Water, Sanitation, and Hygiene behavior and health. With this study, we want to determine whether multi-faceted contextualized and non-contextualized WASH interventions have a differential impact.

OBJECTIVES. The primary objective is to determine the effectiveness of a contextualized and non-contextualized add-on intervention for improving hand washing (HW) behavior. Secondary objectives include the impact on latrine use, health, coverage of HW and latrine infrastructure, quality of life, and cost-effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* All people above 18 years of age.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1500 (Actual)
Dates: Start 2018-04-23 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Change in hand washing behavior | The outcome is measured at baseline, and after 1 and 2 years of intervention. In addition, a measurement will occur 1 year after the intervention has finished to see whether improvements have been maintained.
  The primary outcome is the percentage of households washing hands. The outcome measure will be obtained by means of a self-developed WASH questionnaire, which involves both multiple choice questions and spot checks.
  A household was defined to have correct HW behavior when they: 1) have a HW station available (spot check), 2) have water and soap available at the HW station (spot check), and 3) indicate to wash their hands with water and soap (questionnaire). The analysis will be repeated for each of the critical times. Critical times of interest include: after defecation or using the latrine, before cooking or handling food, before eating, and before feeding a child.

SECONDARY OUTCOMES:
Change in latrine use behavior | The outcome is measured at baseline, and after 1 and 2 years of intervention. In addition, a measurement will occur 1 year after the intervention has finished to see whether improvements have been maintained.
  Latrine use is assessed by means of a self-developed WASH questionnaire, involving both multiple choice questions and spot checks.
  A household is defined to have correct latrine use behavior when: 1) they have a latrine available (spot check), 2) the latrine minimally includes walls, a roof, a door or curtain, and a slab or concrete floor (spot check), 3) the latrine is clean (spot check), 3) they indicate to normally use the latrine when defecating at home (questionnaire), and 4) they indicate to not defecate in the open when they are at home (questionnaire). A similar analysis will be performed for latrine use behavior when people are elsewhere.
Quality of the hand washing infrastructure | The outcome is measured at baseline, and after 1 and 2 years of intervention. In addition, a measurement will occur 1 year after the intervention has finished to see whether improvements have been maintained.
  Hand washing infrastructure is assessed using a self-developed questionnaire and spot checks. The quality of the HW infrastructure is scored based on the type of HW facility (i.e. running water vs. bucket) (spot check), the presence of water and/or soap (spot check), and whether or not the station is always operational (questionnaire).
Change in health | The outcome is measured at baseline, and after 1 and 2 years of intervention. In addition, a measurement will occur 1 year after the intervention has finished to see whether improvements have been maintained.
  Health is assessed using a self-developed health questionnaire. The questionnaire is used to probe the prevalence rates of diarrhea, vomiting, limitations of daily activities, and need for medical care due to diarrheal illness in the past two weeks. The questionnaire also probes about the prevalence rates of hospitalization due to diarrheal illness in the past twelve months. Prevalence is subdivided into people below 5 years of age and people above 5 years of age. In some questions, a distinction was also made between men and women.
Change in EQ-5D-3L | The outcome is measured at baseline, and after 1 and 2 years of intervention. In addition, a measurement will occur 1 year after the intervention has finished to see whether improvements have been maintained.
  The EQ-5D-3L is a validated questionnaire, examining 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. All items are scored on a 3-point Likert scale. Results of the EQ-5D-3L can be used to calculate the quality-adjusted life-year (QALY), a generic measure of disease burden. The QALY will be used to determine the cost-effectiveness of each intervention arm.
Quality of the latrine infrastructure | The outcome is measured at baseline, and after 1 and 2 years of intervention. In addition, a measurement will occur 1 year after the intervention has finished to see whether improvements have been maintained.
  Latrine infrastructure is assessed using a self-developed questionnaire and spot checks. The quality of the latrine infrastructure is scored based on the type of facility (i.e. does it have a roof, a door, etc.) (spot check), the cleanliness (spot check), and the number of people who use the latrine (questionnaire). Information about whether or not the pit has ever been emptied, and how will also be gathered (questionnaire) as this will allow for the measurement of Sustainable Development Goal (SDG) 6 according to the WHO/UNICEF JMP (https://washdata.org/) tools.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanzania Red Cross Society, Kigoma, Tanzania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dockx K, Van Remoortel H, De Buck E, Schelstraete C, Vanderheyden A, Lievens T, Kinyagu JT, Mamuya S, Vandekerckhove P. Effect of Contextualized Versus Non-Contextualized Interventions for Improving Hand Washing, Sanitation, and Health in Rural Tanzania: Study Design of a Cluster Randomized Controlled Trial. Int J Environ Res Public Health. 2019 Jul 15;16(14):2529. doi: 10.3390/ijerph16142529. PMID 31311186
- See also: Related Info — http://www.cebap.org